CLINICAL TRIAL: NCT05440201
Title: Coupling Between Clotting Characteristics in Chronic Hemodialysis Patients and the Hemodialyzer Patency
Acronym: ClotPara
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: UGent_ClotPara
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Bleeding; Coagulation
MeSH Terms: conditions — Hemorrhage; Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First test session (Experimental): For each patient, the anticoagulant Clexane 50IE/kg is administered in the venous line of the dialysis circuit once blood is detected by the dialysis machine.
  Interventions: Other: Amount of anticoagulant Clexane
- Second test session (Experimental): The dosis of Clexane is lowered or increased by 50%, depending on the results of the fiber patency and clotting characteristics of the previous session.
  Interventions: Other: Amount of anticoagulant Clexane
- Third test session (Experimental): The dosis of Clexane is lowered or increased by 50%, depending on the results of the fiber patency and clotting characteristics of the previous session.
  Interventions: Other: Amount of anticoagulant Clexane
- Fourth test session (Experimental): The dosis of Clexane is lowered or increased by 50%, depending on the results of the fiber patency and clotting characteristics of the previous session.
  Interventions: Other: Amount of anticoagulant Clexane

INTERVENTIONS:
Other: Amount of anticoagulant Clexane — Change (increase/decrease) the amount of Clexane administered at the dialysis start.

SUMMARY:
Twenty stable chronic hemodialysis patients are included and will undergo one, two, three or four midweek test dialysis sessions, depending on a flow chart to follow.

All patients are started (week 1) with an anticoagulant Clexane 50IE/kg and are dialyzed with their regular dialyzer and dialysis machine. Depending on the results of measured clotting characteristics and of the dialyzer scanning (i.e. percentage open fibers), it is decided (via the flow chart) whether the patient gets a second session (and so on) with an adapted anticoagulation therapy to ameliorate fiber patency while limiting bleedings.

DETAILED DESCRIPTION:
Twenty stable chronic hemodialysis (HD) patients with a well functioning vascular access will be included. Patients have a hematocrit higher than 30%, and have no known heparin allergy, no severe thrombocytopenia (platelets more than 50.000/µL) or active infection. Patients are not treated with vitamin K antagonists.

The study is limited to maximum four test sessions at midweek per patient. Patients are dialysed with their regular dialyzer on their regular dialysis machine. Patients will get a dialysis of 240min with blood flow 300mL/min and dialysate flow 500mL/min. Ultrafiltration is set according to the patient's needs. As usual, patients will get an administration of an anticoagulant in the dialysis circuit to avoid clotting of the extracorporeal circuit.

At the start of the first test session, patients receive the anticoagulant Clexane 20-30IE/kg (0.2-0.3mg/kg - rounded to 10).

In these 20 patients, clotting characteristics are measured by performing clotting tests, such as thrombin generation test, thrombo-elastogram with Rotem, Platelet Function Analysis (PFA), flow chamber, and the measurement of biochemical markers such as anti-thrombin-III (AT-III), p-selectin, and antiXa. For these measurements, blood is sampled predialysis, 30min after dialysis start, and post dialysis.

In order to link these clotting characteristics with dialyzer patency, the dialyzer will be scanned post dialysis with a gold standard micro Computed Tomography (CT) technique. At the end of the dialysis session, a standard rinsing procedure is applied. The dialyzer is then dried for 12-24 hours by continuous positive pressure ventilation in blood and dialysate compartment. During scanning, the dialyzer is mounted vertically on a rotating disc in front of the X-rays source. After image reconstruction, we get images of cross sections of the dialyzer. The non-blocked fibers are counted with an open source computer program used for biological image analysis. By comparing the number of non-blocked fibers with the total number of fibers in a non-used dialyzer, the percentage of fiber blocking can be derived.

By comparing the percentage of fiber blocking with the clotting characteristics in the patient, insight can be obtained in the value of the different clotting characteristics.

Based on the results of the first midweek session, it is decided (based on a flow chart) whether the patient will also get a second, third and eventual fourth dialysis test session at midweek with an adapted anticoagulation therapy to ameliorate fiber patency while limiting bleedings.

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis patients
* well functioning vascular access
* hematocrit higher than 30%

Exclusion Criteria:

* known heparin allergy
* severe thrombocytopenia (platelets more than 50.000/µL)
* active infection
* treatment with vitamin K antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Dialyzer fiber patency | 4 midweek sessions
  Percentage of open fibers in de dialyzer post dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, Prof dr, Principal Investigator — UZ Gent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No